CLINICAL TRIAL: NCT01285310
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study, To Compare the Efficacy and Safety of Two Doses of Apremilast (CC-10004) in Subjects With Active Rheumatoid Arthritis Who Have Had an Inadequate Response to Methotrexate
Brief Title: Study of Apremilast to Evaluate the Safety and Effectiveness for Patients With Rheumatoid Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study is terminated due to lack of efficacy
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-10004-RA-002; 2010-019926-15 (EudraCT Number)
Record Dates: First submitted 2010-11-19; First posted 2011-01-28 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2020-05-08 (Actual); Status verified 2020-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid, Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Apremilast 30 mg (Experimental)
  Interventions: Drug: Apremilast 30 mg
- Apremilast 20 mg (Experimental)
  Interventions: Drug: Apremilast 20 mg; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apremilast 30 mg — 30 mg oral Apremilast tablets administered twice daily (BID) for 24 weeks during the placebo-controlled phase followed by 30mg Apremilast tablets administered BID for up to 1.5 years in the active treatment / active treatment extension phase.
  Other Names: CC-10004
  Arms: Apremilast 30 mg
Drug: Apremilast 20 mg — 20 mg oral Apremilast tablets administered twice daily (BID) for 24 weeks during the placebo-controlled phase followed by 20mg Apremilast tablets administered BID for up to 1.5 years in the active treatment / active treatment extension phase.
  Arms: Apremilast 20 mg
Drug: Placebo — Oral Placebo tablets administered twice daily (BID) for 24 weeks during the placebo-controlled phase followed by 20mg Apremilast tablets administered BID for up to 1.5 years in active treatment / active treatment extension phase. Participants who are nonresponders will advance early to 20 mg Apremilast BID at Week 16.
  Arms: Apremilast 20 mg; Placebo

SUMMARY:
The purpose of this study is to determine whether Apremilast is safe and effective in the treatment of patients with rheumatoid arthritis, specifically in improving signs and symptoms of rheumatoid arthritis (tender and swollen joints, pain, physical function and structure) in treated patients who have had an inadequate response to Methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Must have a documented diagnosis of Rheumatoid Arthritis (1987 American College of Rheumatology Criteria) with onset of signs/symptoms of disease ≥ 4 months of duration from randomization.
* Must be receiving treatment on an outpatient basis.
* Must have active disease despite current methotrexate treatment as defined below:

  * ≥ 6 swollen joints (66 swollen joint count) AND
  * ≥ 6 tender joints (68 tender joint count)

    -. Must meet at least one of the four lab requirements below:
  * High Sensitivity C-Reactive Protein (hsCRP) ≥ 10 mg/L
  * Erythrocyte Sedimentation Rate (ESR) > 28 mm after the first 1 hour
  * Positive for Rheumatoid Factor (RF)
  * Positive for Anti-cyclic Citrullinated Peptide (anti-CCP) antibodies
* For participants participating in the Magnetic Resonance Imaging (MRI) assessment:

  • Must have Rheumatoid Arthritis joint involvement, as assessed by swollen joint counts in: 1) at least two Metacarpophalangeal (MCP) swollen joints on the same hand, or 2) at least one swollen Metacarpophalangeal (MCP) joint and swollen wrist on the same hand.
* Must have been treated with methotrexate for at least 4 months prior to randomization, and must be on stable dose. Participants will be required to maintain their stable dose through Week 52 of the study. Oral folate (folic acid) supplementation is required with a minimum dose of 5 mg/week, or instead leucovorin may be used up to 10 mg/week orally.

  • Non-steroidal anti-inflammatory drugs (NSAIDs) and pain medications are allowed, however, must be on stable regimen for at least 7 days prior to randomization and through Week 52 of the study.
* Oral corticosteroids (if taken) are allowed, however, must be on stable dose of prednisone ≤ 10 mg/day or equivalent for at least 28 days prior to randomization and through Week 52 of the study.
* Must meet the following laboratory criteria at screening:

  * White blood cell count ≥ 3000/mm^3 (≥ 3.0 x 10^9/L) and < 14,000/mm^3 (< 14 x 10^9/L)
  * Platelet count (≥ 100,000/μL ((≥ 100 x 10^9/L)
  * Serum creatinine ≤ 1.5 mg/dL (≤ 132.6 μmol/L)
  * Aspartate aminotransferase or serum glutamic oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase or serum glutamic-pyruvic transaminase (ALT/ SGPT) ≤ 2 x upper limit of normal (ULN). If initial test shows Aspartate aminotransferase (AST) or alanine aminotransferase (SLT) or 2 times the upper limit of normal (ULN), one repeat test is allowed during the screening period.
  * Total bilirubin ≤ 2 mg/dL (≤ 34 μmol/L). If initial test result is > 2 mg/dL, one repeat test is allowed during the screening period.
  * Hemoglobin ≥ 9 g/dL (≥ 5.6 mmol/L)
  * Hemoglobin A1c ≤ 9.0%
  * Negative for hepatitis B surface antigen
  * Negative for hepatitis C antibody
* Males who engage in activity in which conception is possible must use protocol described barrier contraception while on Investigational Product and for at least 28 days after the last dose of Investigational Product.
* Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline. FCBP who engage in activity in which conception is possible must use protocol described contraception while on Investigational Product and for at least 28 days after taking the last dose or Investigational Product.

Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following randomization.
* Rheumatic autoimmune disease other than Rheumatoid Arthritis, including systemic lupus erythematosus, mixed connective tissue disease, scleroderma, polymyositis or significant systemic involvement secondary to Rheumatoid Arthritis (eg, vasculitis, pulmonary fibrosis or Felty syndrome). Sjögren syndrome secondary to Rheumatoid Arthritis is allowable.
* Functional Class IV as defined by the American College of Rheumatology (ACR) Classification of Functional Status in Rheumatoid Arthritis.
* Prior history of, or current, inflammatory joint disease other than Rheumatoid Arthritis (eg, gout, reactive arthritis, psoriatic arthritis, ankylosing spondylitis, Lyme disease).
* Receiving treatment with Disease-modifying antirheumatic drugs (DMARDs) (other than methotrexate), including biologic Disease-modifying antirheumatic drugs (DMARDs)Previous use is only allowed after adequate washout prior to randomization.
* Inadequate response to treatment with an anti-tumor necrosis factor (anti-TNF) agent. Patients who terminated previous anti-tumor necrosis factor (anti-TNF) treatment due to cost or safety reason, such as discomfort with the subcutaneous injections, may participate in this study after adequate washout.
* Treatment with any investigational agent within four weeks (or five half-lives of the investigational drug, whichever is longer) of screening.
* Previous treatment with any cell depleting therapies, including investigational agents.
* Treatment with intravenous gamma globulin, plasmapheresis or Prosorba® column within 6 months of baseline.
* Intra-articular or parenteral corticosteroids are not allowed within 6 weeks prior to randomization.
* Any previous treatment with alkylating agents such as cyclophosphamide or chlorambucil, or with total lymphoid irradiation.
* Pregnant women or nursing (breast feeding) mothers.
* Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary (including severe or very severe chronic obstructive pulmonary disease), renal, hepatic, endocrine (including uncontrolled diabetes mellitus as defined by Hemoglobin A1c > 9.0%) or gastrointestinal (GI) disease.
* Uncontrolled disease states, such as asthma, psoriasis or inflammatory bowel disease, where flares are commonly treated with oral or parenteral corticosteroids.
* Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections (including but not limited to tuberculosis and atypical mycobacterial disease, Hepatitis B and C, and herpes zoster, but excluding onychomycosis) or any major episode of infection requiring hospitalization or treatment with IV or oral antibiotics within 4 weeks of screening.
* History of positive Human Immunodeficiency Virus (HIV), or congenital or acquired immunodeficiency (eg, Common Variable Immunodeficiency Disease).
* History of malignancy, including solid tumors and hematologic malignancies (except basal cell carcinoma of the skin that has been excised and cured).
* History of alcohol, drug or chemical abuse within the 6 months prior to screening.
* Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
* Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
* Any condition that in the investigator's opinion would interfere significantly with the efficacy evaluations, including the pain and joint assessments (eg, fibromyalgia).

For Magnetic Resonance Imaging (MRI) Only:

* Receiving medication(s) or will require medication(s) during the study that impact on vascular flow (eg, nitrates, calcium channel blockers, ergot containing drugs) on the day of the Magnetic Resonance Imaging (MRI test and in the investigator's judgement the subject cannot hold back from taking these medications on the day of the Magnetic Resonance Imaging (MRI) prior to the Magnetic Resonance Imaging (MRI) test. The subject can continue taking the medication(s) at any time after the Magnetic Resonance Imaging (MRI) test is completed, as clinically indicated and scheduled. Exclusions of antihypertensive and migraine medications can be determined after discussion with the Sponsor.
* Unable to undergo an Magnetic Resonance Imaging (MRI) examination, including but not limited to the presence of a pacemaker, defibrillator, or other implanted device such as anterior interbody cages, aneurysm clip, pedicle screws, or any other metal contained in the body (eg, such as tattoos that contain metallic pigment, or metal in the eyes from metal grinding [eg, a metal worker, etc]), or severe claustrophobia, or any other contraindication to an Magnetic Resonance Imaging (MRI) as per local imaging center guidelines.
* Allergic or adverse reactions to gadolinium
* Estimated glomerular filtration rate (eGFR) below 60 mL/min/1.73m2 (based on the Modification of Diet in Renal Disease [MDRD] formula).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2010-12-09 (Actual); Primary Completion 2012-02-21 (Actual); Study Completion 2012-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (50):
- United States (29):
  - ArthroCare, Arthritis Care Research, Gilbert, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - TriWest Research Associates, La Mesa, California
  - Desert Medical Advances, Palm Desert, California
  - Stanford University Medical Center, Palo Alto, California
  - Med Investigations/Sierra, Roseville, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - Denver Arthritis Clinic, Denver, Colorado
  - In Vivo Clinical Research, Doral, Florida
  - San Marcus Research Clinic, Miami, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Jeffrey Alper, MD Research, Naples, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Tampa Medical Group, PA, Tampa, Florida
  - Alastair Kennedy, MD, Vero Beach, Florida
  - LaPorte County Institute for Clinical Research, Inc., Michigan City, Indiana
  - Associated Internal Medicine Specialists, PC, Battle Creek, Michigan
  - Saint Paul Rheumatology, Eagan, Minnesota
  - Physician's East, Greenville, North Carolina
  - David R. Mandel, M.D., Inc., Mayfield, Ohio
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Austin Regional Clinic, Austin, Texas
  - Metroplex Research Center, Dallas, Texas
  - Modern Research Associates, Dallas, Texas
  - Sun Research Institute, San Antonio, Texas
  - Stone Oak Rheumatology, San Antonio, Texas
  - Center for Excellence in Aging and Geriatric Health, Williamsburg, Virginia
  - Arthritis Northwest, Rheumatology, Spokane, Washington
- Czechia (7):
  - Revmatologie s.r.o., Brno
  - L.K.N. Arthrocentrum s.r.o., Hlučín
  - ARTMEDI UPD s.r.o., Hostivice
  - Revmatologicky ustav, Prague
  - Revmatologicka ambulance, Prague
  - Fakultni Thomayerova nemocnice s poliklinikou, Prague
  - PV - MEDICAL, s.r.o., Zlín
- Poland (10):
  - NZOZ Osteo-Medic s.c. Artur Racewicz, Jerzy Supronik, Bialystok
  - NZOZ Centrum Osteoporozy i Chorob Kostno-Stawowych, Bialystok
  - Szpital Uniwersytecki nr 2 im. Dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Centrum Kliniczno-Badawcze, Elblag
  - Centrum Leczenia Chorob Cywilizacyjnych, Gdynia
  - Centrum Leczenia Chorob Cywilizacyjnych, Katowice
  - Malopolskie Centrum Medyczne (408), Krakow
  - Niepubliczny Zaklad Opieki Zdrowotnej REUMED, Lublin
  - Prywatna Praktyka Lekarska Pawel Hrycaj, Poznan
  - Centrum Leczenia Chorob Cywilizacyjnych, Warsaw
- Spain (4):
  - Hospital Universitario a Coruña, A Coruña
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
  - Hospital Sierrallana, Torrelavega

REFERENCES:
- [Derived] Genovese MC, Jarosova K, Cieslak D, Alper J, Kivitz A, Hough DR, Maes P, Pineda L, Chen M, Zaidi F. Apremilast in Patients With Active Rheumatoid Arthritis: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study. Arthritis Rheumatol. 2015 Jul;67(7):1703-10. doi: 10.1002/art.39120. PMID 25779750

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 302 subjects were screened for inclusion in this study, and 237 participants randomized in parallel in a 1:1:1 ratio to treatment groups. The first participant was enrolled on 27 December 2010; the last participant completed week 24 visit on 23 February 2012.
Groups:
- Placebo: Participants initially randomized to placebo tablets twice daily in the 24-week placebo-controlled phase. Participants who did not have at least 20% improvement in swollen and tender joint counts at Week 16 were transitioned onto 20 mg Apremilast twice daily (early escape), and were designated as Placebo/Apremilast 20mg EE.
- Apremilast 20 mg: Participants initially randomized to receive 20 mg apremilast tablets twice daily in the 24-week placebo-controlled phase and continued to receive 20 mg apremilast tablets twice daily (BID) for up to Week 52 in the active treatment.
  At week 52, participants were given the option to remain on active treatment for 1 additional year (extension phase) as assigned during the active treatment phase.
- Apremilast 30 mg: Participants initially randomized to receive 30 mg apremilast tablets twice daily in the 24-week placebo-controlled phase and continued to receive 30 mg apremilast tablets twice daily (BID) for up to Week 52 in the active treatment.
  At week 52, participants were given the option to remain on active treatment for 1 additional year (extension phase) as assigned during the active treatment phase.
- Placebo/Apremilast 20mg EE: Participants initially randomized to receive placebo twice daily and were transitioned due to early escape (EE) at Week 16 to receive 20 mg apremilast for up to week 24.
  At week 24, participants were continued on Apremilast 20 mg BID for up to Week 52.
  At week 52, they were given the option to remain on active treatment for 1 additional year (extension phase) as assigned during the active treatment phase.
- Placebo / Apremilast 20 mg XO: Participants initially randomized to receive placebo twice daily who were transitioned at Week 24 (XO) to receive 20 mg apremilast for up to Week 52.
  At week 52, they were given the option to remain on active treatment for 1 additional year (extension phase) as assigned during the active treatment phase.
Period: Placebo Controlled Phase: Weeks 0-24
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo/Apremilast 20mg EE | Placebo / Apremilast 20 mg XO
Started | 79 | 82 | 76 | 0 | 0
Completed | 70 (1 participant chose not to enter the active treatment phase) | 67 (Four participants chose not to enter the active treatment phase) | 61 (1 participant chose not to enter active treatment phase) | 0 | 0
Not Completed | 9 | 15 | 15 | 0 | 0
Not completed — Adverse Event | 3 | 4 | 6 | 0 | 0
Not completed — Lack of Efficacy | 1 | 7 | 3 | 0 | 0
Not completed — Non-compliance | 1 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0
Not completed — Other | 1 | 0 | 1 | 0 | 0
Period: Active Treatment Phase: Weeks 25-52
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo/Apremilast 20mg EE | Placebo / Apremilast 20 mg XO
Started | 0 | 63 | 60 | 27 | 42
Completed | 0 | 31 | 34 | 17 | 23
Not Completed | 0 | 32 | 26 | 10 | 19
Not completed — Adverse Event | 0 | 2 | 3 | 0 | 2
Not completed — Lack of Efficacy | 0 | 4 | 3 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 2 | 2
Not completed — Study Termination by sponsor | 0 | 21 | 19 | 6 | 15
Not completed — Other | 0 | 1 | 0 | 0 | 0
Not completed — Non-compliance | 0 | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) The FAS consisted of all participants who were randomized as specified per protocol during the placebo controlled period.
Groups:
- Placebo: Placebo: Oral Placebo tablets administered twice daily (BID) for 24 weeks during the placebo-controlled phase followed by 20mg Apremilast tablets administered BID for up to 1.5 years in active treatment / active treatment extension phase. Participants who are nonresponders were transitioned early to 20 mg Apremilast BID at Week 16.
- Apremilast 20 mg: Apremilast 20 mg: 20 mg oral Apremilast tablets administered twice daily (BID) for 24 weeks during the placebo-controlled phase and continued 20mg Apremilast tablets administered BID for up to 1.5 years in the active treatment / active treatment extension phase.
- Apremilast 30 mg: Apremilast 30 mg: 30 mg oral Apremilast tablets administered twice daily (BID) for 24 weeks during the placebo-controlled phase and continued 30mg Apremilast tablets administered BID for up to 1.5 years in the active treatment / active treatment extension phase.
- Total: Total of all reporting groups
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Total
Number analyzed (Participants) | 79 | 82 | 76 | 237
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (12.45) | 58.6 (11.84) | 52.6 (11.87) | 56.0 (12.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 65 | 55 | 182
  Male | 17 | 17 | 21 | 55
Duration of Rheumatoid Arthritis Diagnosis [Mean (Standard Deviation); unit: years] | 11.98 (12.104) | 8.46 (6.856) | 7.76 (7.833) | 9.41 (9.351)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 20% Improvement (ACR 20) Response at Week 16
Description: Percentage of participants with an American College of Rheumatology 20% Improvement (ACR 20) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met:
  * ≥ 20% improvement in 68 tender joint count;
  * ≥ 20% improvement in 66 swollen joint count; and
  * ≥ 20% improvement in at least 3 of the 5 following parameters: Subject's assessment of pain (measured on a 100 mm visual analog scale [VAS]); Subject's global assessment of disease activity (measured on a 100 mm VAS); Physician's global assessment of disease activity (measured on a 100 mm VAS); Subject's self-assessment of physical function (Health Assessment Questionnaire - Disability Index ([HAQ-DI]); C-Reactive Protein.
Time Frame: Baseline and Week 16
Population: Full analysis set consisting of all participants randomized as specified in the protocol; participants who were randomized in error and did not receive any dose of study drug were excluded. Participants who withdrew early or who did not have sufficient data for a definitive determination of response status at Week 16 were counted as non-responders.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants initially randomized to receive placebo tablets twice daily.
- Apremilast 20 mg: Participants initially randomized to receive 20 mg apremilast tablets twice daily.
- Apremilast 30 mg: Participants initially randomized to receive 30 mg apremilast tablets twice daily.
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 79 | 82 | 76
percentage of participants | 35.4 | 28 [-27.7 to 7.0] | 34.2 [-16.2 to 13.8]
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Significance testing was done using the following closed procedure; if the overall test among treatments is statistically significant at the 0.05 level, pair-wise comparisons (30 mg versus PBO, and 20 mg versus PBO, using a 0.05 two-sided significance level) will be performed; Test type: Superiority or Other; p = 0.3134, Chi-squared; Risk Difference (RD) = -7.4, 95% CI 2-sided [-27.1 to 7.0] — 2-sided 95% CI of the proportion difference is based on a normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p = 0.8721, Chi-squared; Risk Difference (RD) = -1.2, 95% CI 2-sided [-16.2 to 13.8] — 2-sided 95% CI is based on a normal approximation to the binomial distribution

2. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 16
Description: The Health Assessment Questionnaire - Disability Index (HAQ-DI) was a patient-reported questionnaire consisting of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and usual activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task are summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. Negative mean changes from Baseline in the overall score indicate improvement in functional ability.
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline value and at least 1 post-baseline value at or prior to Week 16 are included; Last observation carried forward (LOCF) imputation was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 78 | 80 | 76
units on a scale | -0.106 (0.4173) | -0.114 (0.5036) | -0.209 (0.4469)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = -0.004 — Based on an analysis of covariance model for the change from baseline at Week 16, with treatment group as a factor and the baseline value as a covariate
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS Mean Difference = -0.091 — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 20% Improvement (ACR 20) Response at Week 24
Description: as for outcome 1
Time Frame: Baseline and Week 24
Population: Full analysis set; Participants who discontinued early, escaped early at Week 16 or who did not have sufficient data for a definitive determination of response status at Week 24 were counted as non-responders.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants initially randomized to receive placebo tablets twice daily. Participants who did not have at least 20% improvement in swollen and tender joint counts at Week 16 were transitioned onto 20 mg apremilast twice daily (early escape) and were designated as Placebo/Apremilast 20mg EE.
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 79 | 82 | 76
percentage of participants | 24.1 | 19.5 | 27.6
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Risk Difference (RD) = -4.5
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Risk Difference (RD) = 3.6

4. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) at Week 24
Description: The Health Assessment Questionnaire - Disability Index (HAQ-DI) is a patient-reported questionnaire consisting of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and usual activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task are summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. Negative mean changes from Baseline in the overall score indicate improvement in functional ability.
Time Frame: Baseline and Week 24
Population: Full analysis set; participants with a baseline value and at least 1 post-baseline value at or prior to Week 24 are included; LOCF imputation was used. The Week 16 value was carried over to Week 24 for participants who escaped early at Week 16.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 78 | 80 | 76
units on a scale | -0.069 (0.4328) | -0.080 (0.4653) | -0.227 (0.4910)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Based on an analysis of covariance model for the change from baseline at Week 24; treatment group as a factor and the baseline value as a covariate; LS Mean Difference = -0.007
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Least Squares Mean Difference = -0.150 — Based on an analysis of covariance model for the change from baseline at Week 24, treatment group as a factor and the baseline value as a covariate

5. Secondary Outcome: Change From Baseline in the Medical Outcome Study Short Form 36-item (SF-36) Physical Functioning Domain at Week 16
Description: The Medical Outcome Study Short Form 36-Item Health Survey, Version 2 (SF-36) is a self-administered instrument that measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). The concepts measured by the SF-36 are not specific to any age, disease, or treatment group, allowing comparison of relative burden of different diseases and the relative benefit of different treatments. Norm-based scores were used in analyses, calibrated so that 50 is the average score and the standard deviation equals 10. Higher scores indicate a higher level of functioning. The physical functioning domain assesses limitations in physical activities because of health problems. A positive change from baseline score indicates an improvement.
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline value and at least 1 post-baseline value at or prior to Week 16 are included; LOCF imputation was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 78 | 78 | 75
units on a scale | 1.48 (6.937) | 1.64 (7.036) | 3.33 (6.970)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = -0.17 — Based on an analysis of covariance model for the change from baseline at Week 16; treatment group as a factor and the baseline value as a covariate
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS Mean Difference = 1.77 — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Change From Baseline in the Clinical Disease Activity Index (CDAI) at Week 16
Description: The Clinical Disease Activity Index (CDAI) is a composite index that is calculated as the sum of the:
  * 28 tender joint count (TJC),
  * 28 swollen joint count (SJC),
  * Subject's Global Assessment of Disease Activity measured on a 100 mm visual analog scale (VAS), where 0 mm = lowest disease activity and 100 mm = highest;
  * Physician's Global Assessment of Disease Activity -measured on a 100 mm VAS, where 0 mm = lowest disease activity and 100 mm = highest.
  The CDAI score ranges from 0-76 where lower scores indicate less disease activity. The following thresholds of disease activity have been defined for the CDAI:
  Remission: ≤ 2.8; Low Disease Activity: > 2.8 and ≤ 10; Moderate Disease Activity: > 10 and ≤ 22; High Disease Activity: > 22
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline value and at least 1 post-baseline value at or prior to Week 16 are included. LOCF imputation was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 77 | 79 | 76
units on a scale | -11.52 (14.850) | -9.49 (12.998) | -11.38 (13.230)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Based on an analysis of covariance model for the change from baseline at Week 16; treatment group as a factor and the baseline value as a covariate; LS Mean Difference = 1.21
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.70

7. Secondary Outcome: Percentage of Participants Who Achieve Low Disease Activity or Remission Based on the Clinical Disease Activity Index (CDAI) ≤ 10 at Week 16
Description: as for outcome 6
Time Frame: Baseline and Week 16
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 79 | 82 | 76
percentage of participants | 17.7 | 12.2 | 10.5
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Risk Difference (RD) = -5.5
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Risk Difference (RD) = -7.2

8. Secondary Outcome: Change From Baseline in Disease Activity Score 28 (DAS28) (Using C-Reactive Protein) (CRP) at Week 16
Description: The DAS28 measures the severity of disease at a specific time and is derived from the following variables:
  * 28 tender joint count (TJC28)
  * 28 swollen joint count (SJC28), which do not include the distal interphalangeal (DIP) joints, the hip joint, or the joints below the knee;
  * C-reactive protein (CRP)
  * Subject's global assessment of disease activity (SGA )
  DAS28 values range from 2.0 to 10.0 while higher values mean a higher disease activity.
  A DAS28 score higher than 5.1 indicates high disease activity, a DAS28 score less than 3.2 indicates low disease activity, and a DAS28 score less than 2.6 indicates clinical remission.
Time Frame: Baseline and Week 16
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 78 | 80 | 76
units on a scale | -0.90 (1.272) | -0.73 (1.079) | -0.90 (1.168)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Based on an analysis of covariance model for the change from baseline at Week 16, treatment group as a factor and the baseline value as a covariate; LS Mean Difference = 0.14
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; [statistical method as in outcome 4, analysis 1]; Least Square Mean Difference = -0.02

9. Secondary Outcome: Percentage Change From Baseline in the Tender Joint Count at Week 16
Description: Joint tenderness is the presence of pain in a joint when pressure is applied by the examiner to elicit tenderness. The 68 tender joint count evaluates the following joints: upper-temporomandibular, sternoclavicular, acromioclavicular, shoulder, elbow, wrist, meta-carpophalangeal, proximal interphalangeal and distal interphalangeal; lower: hip, knee, ankle, midtarsal, metatarsophalangeal and proximal interphalangeal.
Time Frame: Baseline and Week 16
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 78 | 81 | 76
percent change | -33.08 (5.154) | -26.92 (5.058) | -33.68 (5.221)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = 6.15 — Based on an analysis of covariance model (Ancova) for the change from baseline at Week 16, with treatment group as a factor and the baseline value as a covariate
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS Mean Difference = -0.61 — [estimate comment as in outcome 9, analysis 1]

10. Secondary Outcome: Percentage Change From Baseline in the Swollen Joint Count at Week 16
Description: Joint swelling is soft tissue swelling that is detectable along the joint margins and is assessed by inspection and direct palpation of the joint, by the examiner. The ACR 66 swollen joint count evaluates the following joints: upper-temporomandibular, sternoclavicular, acromioclavicular, shoulder, elbow, wrist, metacarpophalangeal, proximal interphalangeal and distal interphalangeal; lower: knee, ankle, midtarsal, metatarsophalangeal and proximal interphalangeal.
Time Frame: Baseline and Week 16
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 78 | 81 | 76
percent change | -36.96 (5.432) | -34.38 (5.328) | -40.22 (5.502)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = 2.58 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS Mean Difference = -3.26

11. Secondary Outcome: Percentage Change From Baseline in the Subject Assessment of Pain at Week 16
Description: The Subject Assessment of Pain was measured asking the participant to place a vertical line on a 100-mm visual analog scale on which the left-hand boundary (score = 0 mm) represents "no pain," and the right-hand boundary (score = 100 mm) represents "pain as severe as can be imagined." The distance from the mark to the left-hand boundary was recorded in millimeters.
Time Frame: Baseline and Week 16
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 78 | 80 | 76
percent change | 30.50 (16.584) | -5.03 (16.369) | -7.87 (16.800)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Difference in LS Means = -35.54 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Difference in LS Means = -38.37 — [estimate comment as in outcome 2, analysis 1]

12. Secondary Outcome: Percentage Change From Baseline in the Subject Global Assessment of Disease Activity at Week 16
Description: The Subject Global Assessment of Disease Activity was measured asking the participant to place a vertical line on a 100-mm visual analog scale on which the left-hand boundary (score = 0 mm) represents " lowest disease activity," and the right-hand boundary (score = 100 mm) represents " highest disease activity." The distance from the mark to the left-hand boundary was recorded in millimeters.
Time Frame: Baseline and Week 16
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 79 | 82 | 76
percent change | 10.84 (10.004) | -3.50 (9.872) | 11.19 (10.131)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Difference in LS Means = -14.35 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Difference in LS Means = 0.34 — [estimate comment as in outcome 2, analysis 1]

13. Secondary Outcome: Percentage Change From Baseline in the Physician Global Assessment of Disease Activity at Week 16
Description: The Physician Global Assessment of Disease Activity was measured asking the physician to assess the subject's current arthritis disease activity by placing a vertical line on a 100-mm visual analog scale on which the left-hand boundary (score = 0 mm) represents " lowest disease activity," and the right-hand boundary (score = 100 mm) represents " highest disease activity." The distance from the mark to the left-hand boundary was recorded in millimeters.
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 77 | 80 | 76
percent change | -28.82 (4.478) | -28.22 (4.440) | -32.66 (4.540)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Difference in LS Means = 0.59 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Difference in LS Means = -3.84 — [estimate comment as in outcome 2, analysis 1]

14. Secondary Outcome: Percentage Change From Baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Week 16
Description: as for outcome 2
Time Frame: Baseline and Week 16
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 78 | 80 | 76
percent change | -9.43 (5.307) | -3.50 (5.234) | -10.20 (5.416)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Difference in LS Means = 5.93 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Difference in LS Means = -0.77 — [estimate comment as in outcome 2, analysis 1]

15. Secondary Outcome: Percentage Change From Baseline in the High Sensitivity C-Reactive Protein (CRP) at Week 16
Description: C-Reactive Protein (CRP) is a substance produced by the liver that increases in the presence of inflammation in the body. An elevated CRP level is identified with blood tests and is considered a non-specific "marker" for disease.
Time Frame: Baseline and Week 16
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 78 | 81 | 76
percent change | 41.99 (30.559) | 46.69 (30.027) | 100.04 (31.127)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Difference in LS Means = 4.70 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Difference in LS Means = 58.05

16. Secondary Outcome: Percentage Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Week 16
Description: The erythrocyte sedimentation rate (ESR) is a blood test that can reveal inflammatory activity. The subject's blood is placed in a tall, thin tube, red erythrocytes gradually settle to the bottom. Inflammation can cause the cells to clump together. Because these clumps of cells are denser than individual cells, they settle to the bottom more quickly.
  The ESR test measures the distance red blood cells fall in a test tube in one hour. The farther the red blood cells have descended, the greater the inflammatory response.
Time Frame: Baseline and Week 16
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 78 | 81 | 76
percent change | 6.81 (10.633) | 13.98 (10.522) | -9.39 (10.681)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Difference in LS Means = 7.18 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Difference in LS Means = -16.19 — [estimate comment as in outcome 2, analysis 1]

17. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score at Week 16
Description: The FACIT-Fatigue scale was a 13-item self-administered questionnaire that assesses both the physical and functional consequences of fatigue. Each question is answered on a 5-point scale, where 0 means "not at all," and 4 means "very much." The FACIT-Fatigue scale score ranges from 0 to 52, with higher scores denoting lower levels of fatigue.
  A positive change from baseline score indicates an improvement.
Time Frame: Baseline and Week 16
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 78 | 78 | 75
units on a scale | 2.7 (0.96) | 1.5 (0.96) | 2.6 (0.98)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = -1.2 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Least Square Mean Difference = -0.1 — [estimate comment as in outcome 2, analysis 1]

18. Secondary Outcome: Percentage of Participants Who Achieve an Improvement of ≥ 0.22 Units From Baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 16
Description: as for outcome 2
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 79 | 82 | 76
percentage of participants | 39.2 | 35.4 | 52.6
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Risk Difference (RD) = -3.9
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Risk Difference (RD) = 13.4

19. Secondary Outcome: Percentage of Participants Who Achieve an Improvement of at Least 4 Units From Baseline in the Functional Assessment of Chronic Illness Therapy -Fatigue (FACIT-Fatigue) at Week 16
Description: as for outcome 17
Time Frame: Baseline and Week 16
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Groups:
- Apremilast 20 mg: .Participants initially randomized to receive 20 mg apremilast tablets twice daily.
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 79 | 82 | 76
percentage of participants | 39.2 | 35.4 | 42.1
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Risk Difference (RD) = -3.9
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Risk Difference (RD) = 2.9

20. Secondary Outcome: Percentage of Participants Who Achieve the European League Against Rheumatism (EULAR) Response Criteria Using CRP at Week 16
Description: EULAR response criteria classify each participant as a good, moderate or non-responder to treatment based on the degree of improvement from baseline and the level of disease activity at the endpoint. EULAR response is derived using the individual subject's DAS28 as the measure of severity of disease.
  Good or moderate response is defined as follows: Good response: DAS28 at the time point ≤ 3.2 and improvement from baseline > 1.2 Moderate response: DAS28 at the time point > 3.2 and improvement from baseline > 1.2, or DAS28 at the time point ≤ 5.1 and improvement from baseline > 0.6 and ≤ 1.2
Time Frame: Baseline and Week 16
Population: Full analysis set; Participants who discontinued early, or who did not have sufficient data for a definitive determination of response status at Week 16 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 79 | 82 | 76
percentage of participants | 46.8 | 41.5 | 44.7
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Risk Difference (RD) = -5.4
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Risk Difference (RD) = 2.1

21. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 50% Improvement (ACR 50) Response at Week 16
Description: Percentage of participants with an American College of Rheumatology 50% Improvement (ACR50) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met:
  * ≥ 50% improvement in 68 tender joint count;
  * ≥ 50% improvement in 66 swollen joint count; and
  * ≥ 50% improvement in at least 3 of the 5 following parameters:
  Subject's assessment of pain (measured on a 100 mm visual analog scale [VAS]); Subject's global assessment of disease activity (measured on a 100 mm VAS); Physician's global assessment of disease activity (measured on a 100 mm VAS); Subject's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [(HAQ-DI)]); C-Reactive Protein.
Time Frame: Baseline and Week 16
Population: as for outcome 20
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 79 | 82 | 76
percentage of participants | 11.4 | 4.9 | 9.2
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Risk Difference (RD) = -6.5
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Risk Difference (RD) = -2.2

22. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 70% Improvement (ACR 70) Response at Week 16
Description: Percentage of participants with an American College of Rheumatology 70% Improvement (ACR70) response. A participant was a responder if the following 3 criteria for improvement from baseline were met:
  * ≥ 70% improvement in 68 tender joint count;
  * ≥ 70% improvement in 66 swollen joint count; and
  * ≥ 70% improvement in at least 3 of the 5 following parameters: Subject's assessment of pain (measured on a 100 mm visual analog scale [VAS]); Subject's global assessment of disease activity (measured on a 100 mm VAS); Physician's global assessment of disease activity (measured on a 100 mm VAS); Subject's self-assessment of physical function (Health Assessment Questionnaire - Disability Index ([HAQ-DI]); C-Reactive Protein
Time Frame: Baseline and Week 16
Population: Full Analysis Set = The FAS consisted of all participants who were randomized as specified per protocol during the placebo controlled period. The last observed joint assessment (at baseline or post-baseline) was used for joints unassessed at Week 16.
Measure: Number; unit: percent of participants
Groups:
- Placebo: Participants initially randomized to receive placebo tablets twice daily. Participants who did not have at least 20% improvement in swollen and tender joint counts at Week 16 were transitioned onto 20 mg apremilast twice daily (early escape).
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 79 | 82 | 76
percent of participants | 2.5 | 1.2 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Risk Difference (RD) = -1.3
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Risk Difference (RD) = -2.5

23. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 50% Improvement (ACR 50) Response at Week 24
Description: Percentage of participants with an American College of Rheumatology 50% Improvement (ACR 50) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met:
  * ≥ 50% improvement in 68 tender joint count;
  * ≥ 50% improvement in 66 swollen joint count; and
  * ≥ 50% improvement in at least 3 of the 5 following parameters:
  Subject's assessment of pain (measured on a 100 mm visual analog scale [VAS]); Subject's global assessment of disease activity (measured on a 100 mm VAS); Physician's global assessment of disease activity (measured on a 100 mm VAS); Subject's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [(HAQ-DI)]); C-Reactive Protein.
Time Frame: Baseline and Week 24
Population: Full Analysis Set = The FAS consisted of all participants who were randomized as specified per protocol during the placebo controlled period. The last observed joint assessment (at baseline or post-baseline) was used for joints unassessed at Week 24.
Measure: Number; unit: percentage of participants
Groups:
- Apremilast 30 mg: .Participants initially randomized to receive 30 mg apremilast tablets twice daily
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 79 | 82 | 76
percentage of participants | 6.3 | 4.9 | 15.8
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Risk Difference (RD) = -1.5
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Risk Difference (RD) = 9.5

24. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 70% Improvement (ACR 70) Response at Week 24
Description: Percentage of participants with an American College of Rheumatology 70% Improvement (ACR 70) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met:
  * ≥ 70% improvement in 68 tender joint count;
  * ≥ 70% improvement in 66 swollen joint count; and
  * ≥ 70% improvement in at least 3 of the 5 following parameters:
  Subject's assessment of pain (measured on a 100 mm visual analog scale [VAS]); Subject's global assessment of disease activity (measured on a 100 mm VAS); Physician's global assessment of disease activity (measured on a 100 mm VAS); Subject's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [(HAQ-DI)]); C-Reactive Protein.
Time Frame: Baseline and Week 24
Population: as for outcome 23
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 79 | 82 | 76
percentage of participants | 3.8 | 2.4 | 5.3
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Risk Difference (RD) = -1.4
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Risk Difference (RD) = 1.5

25. Secondary Outcome: Change From Baseline in the Medical Outcome Study Short Form 36-item (SF-36) Physical Functioning Domain at Week 24
Description: The Medical Outcome Study Short Form 36-Item Health Survey, Version 2 (SF-36) is a self-administered instrument that measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). Norm-based scores were used in analyses, calibrated so that 50 is the average score and the standard deviation equals 10. Higher scores indicate a higher level of functioning. The physical functioning domain assesses limitations in physical activities because of health problems. A positive change from Baseline score indicates an improvement.
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Participants initially randomized to receive placebo tablets twice daily. Participants who did not have at least 20% improvement in swollen and tender joint counts at Week 16 were transitioned onto 20 mg apremilast twice daily (early escape) and were designated as Placebo/Apremilast 20mg EE ..
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 78 | 78 | 75
units on a scale | 1.78 (0.849) | 1.66 (0.850) | 3.76 (0.865)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = -0.12 — Based on an analysis of covariance model for the change from baseline at Week 24 with treatment group as a factor and the baseline value as a covariate
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS Mean Difference = 1.98 — [estimate comment as in outcome 25, analysis 1]

26. Secondary Outcome: Change From Baseline in the Clinical Disease Activity Index (CDAI) at Week 24
Description: The Clinical Disease Activity Index (CDAI) is a composite index that is calculated as the sum of the:
  * 28 tender joint count (TJC),
  * 28 swollen joint count (SJC),
  * Subject's Global Assessment of Disease Activity measured on a 100 mm visual analog scale (VAS), where 0 mm = lowest disease activity and 100 mm = highest;
  * Physician's Global Assessment of Disease Activity -measured on a 100 mm VAS, where 0 mm = lowest disease activity and 100 mm = highest.
  The CDAI score ranges from 0-76 where lower scores indicate less disease activity.The following thresholds of disease activity have been defined for the CDAI:
  Remission: ≤ 2.8; Low Disease Activity: > 2.8 and ≤ 10; Moderate Disease Activity: > 10 and ≤ 22; High Disease Activity: > 22
Time Frame: Baseline and Week 24
Population: Full analysis set; Participants who discontinued early, escaped early at Week 16 or who did not have sufficient data for a definitive determination of response status at Week 24 were counted as non-responders. LOCF imputation was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 77 | 79 | 76
units on a scale | -10.40 (1.597) | -9.46 (1.571) | -11.63 (1.602)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = 0.94
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; [statistical method as in outcome 4, analysis 1]; Least Square Mean Difference = -1.24

27. Secondary Outcome: Percentage of Participants Who Achieve Low Disease Activity or Remission Based on the Clinical Disease Activity Index (CDAI) ≤ 10 at Week 24
Description: as for outcome 26
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 79 | 82 | 76
percentage of participants | 16.5 | 12.2 | 21.1
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Difference in proportions = -4.3
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Difference in proportions = 4.6

28. Secondary Outcome: Change From Baseline in Disease Activity Score 28 (DAS28) Using CRP at Week 24
Description: The DAS28 measures the severity of disease at a specific time and is derived from the following variables:
  * 28 tender joint count
  * 28 swollen joint count, which do not include the DIP joints, the hip joint, or the joints below the knee;
  * C-reactive protein (CRP)
  * Subject's Global Assessment of Disease Activity.
  DAS28 values range from 2.0 to 10.0 while higher values mean a higher disease activity.
  A DAS28 score higher than 5.1 indicates high disease activity, a DAS28 score less than 3.2 indicates low disease activity, and a DAS28 score less than 2.6 indicates clinical remission.
Time Frame: Baseline and Week 24
Population: as for outcome 26
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 78 | 80 | 76
units on a scale | -0.82 (0.139) | -0.78 (0.137) | -0.91 (0.141)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = 0.03 — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS Mean Difference = -0.09 — [estimate comment as in outcome 25, analysis 1]

29. Secondary Outcome: Percentage Change From Baseline in the Tender Joint Count at Week 24
Description: as for outcome 9
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 78 | 81 | 76
percent change | -30.81 (5.909) | -26.21 (5.800) | -27.80 (5.987)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = 4.60 — Based on an analysis of covariance model for the change from baseline at Week 24, with treatment group as a factor and the baseline value as a covariate
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS Mean Difference = 3.01 — Based on an analysis of covariance model for the change from baseline at Week 24; treatment group as a factor and the baseline value as a covariate

30. Secondary Outcome: Percentage Change From Baseline in the Swollen Joint Count at Week 24
Description: as for outcome 10
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 78 | 81 | 76
percent change | -34.41 (5.876) | -32.56 (5.764) | -41.43 (5.952)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = 1.86 — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Difference in LS Means = -7.02 — [estimate comment as in outcome 29, analysis 1]

31. Secondary Outcome: Percentage Change From Baseline in the Subject Assessment of Pain at Week 24
Description: as for outcome 11
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 78 | 80 | 76
percent change | 28.16 (16.111) | -6.66 (15.902) | -9.66 (16.320)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = -34.82 — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Difference in LS Means = -37.82 — [estimate comment as in outcome 29, analysis 1]

32. Secondary Outcome: Percentage Change From Baseline in the Subject Global Assessment of Disease Activity at Week 24
Description: as for outcome 12
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 78 | 80 | 76
percent change | 15.04 (8.566) | 0.70 (8.453) | 2.54 (8.675)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Difference in LS Means = -14.34 — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Difference in LS Means = -12.50 — [estimate comment as in outcome 29, analysis 1]

33. Secondary Outcome: Percentage Change From Baseline in the Physician Global Assessment of Disease Activity at Week 24
Description: as for outcome 13
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 77 | 80 | 76
percent change | -29.98 (4.740) | -24.13 (4.700) | -31.78 (4.805)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Difference in LS Means = 5.85 — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Difference in LS Means = -1.80 — [estimate comment as in outcome 29, analysis 1]

34. Secondary Outcome: Percentage Change From Baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Week 24
Description: as for outcome 2
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Placebo: Participants initially randomized to receive placebo tablets twice daily. Participants who did not have at least 20% improvement in swollen and tender joint counts at Week 16 were transitioned onto 20 mg apremilast twice daily (early escape)and were designated as Placebo/Apremilast 20mg EE.
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 78 | 80 | 76
percent change | -6.59 (5.171) | -5.01 (5.100) | -12.30 (5.277)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Difference in LS Means = 1.57 — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Difference in LS Means = -5.72 — [estimate comment as in outcome 29, analysis 1]

35. Secondary Outcome: Percentage Change From Baseline in the High Sensitivity C-Reactive Protein (CRP) at Week 24
Description: as for outcome 15
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 78 | 81 | 76
percent change | 39.14 (30.504) | 47.43 (29.972) | 106.22 (31.071)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Difference in LS Means = 8.29 — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Difference in LS Means = 67.09 — [estimate comment as in outcome 29, analysis 1]

36. Secondary Outcome: Percentage Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Week 24
Description: as for outcome 16
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 78 | 81 | 76
percent change | -0.06 (9.531) | 11.99 (9.431) | -6.60 (9.573)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Difference in LS Means = 12.05 — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Difference in LS Means = -6.54 — [estimate comment as in outcome 29, analysis 1]

37. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score at Week 24
Description: as for outcome 17
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Participants initially randomized to receive placebo tablets twice daily. Participants who did not have at least 20% improvement in swollen and tender joint counts at Week 16 were transitioned to 20 mg apremilast twice daily (early escape) and were designated as Placebo/Apremilast 20mg EE.
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 78 | 78 | 75
units on a scale | 1.7 (1.01) | 0.5 (1.01) | 3.4 (1.03)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = -1.2 — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS Mean Difference = 1.7 — [estimate comment as in outcome 29, analysis 1]

38. Secondary Outcome: Percentage of Participants Who Achieve an Improvement of ≥ 0.22 Units From Baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 24
Description: as for outcome 4
Time Frame: Baseline and Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 79 | 82 | 76
percentage of participants | 20.3 | 25.6 | 32.9
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Risk Difference (RD) = 5.4
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Risk Difference (RD) = 12.6

39. Secondary Outcome: Percentage of Participants Who Achieve an Improvement of at Least 4 Units From Baseline in the Functional Assessment of Chronic Illness Therapy -Fatigue (FACIT-Fatigue) at Week 24
Description: The FACIT-Fatigue scale is a 13-item self-administered questionnaire that assesses both the physical and functional consequences of fatigue. Each question is answered on a 5-point scale, where 0 means "not at all," and 4 means "very much." The FACIT-Fatigue scale score ranges from 0 to 52, with higher scores denoting lower levels of fatigue.
  A positive change from baseline score indicates an improvement.
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 79 | 82 | 76
percentage of participants | 26.6 | 14.6 | 26.3
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Risk Difference (RD) = -11.9
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Risk Difference (RD) = -0.3

40. Secondary Outcome: Percentage of Participants Who Achieve the European League Against Rheumatism (EULAR) Response Criteria Using CRP at Week 24
Description: as for outcome 20
Time Frame: Baseline and Week 24
Population: as for outcome 20
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 79 | 82 | 76
percentage of participants | 40.5 | 29.3 | 35.5
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Risk Difference (RD) = -11.2
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Risk Difference (RD) = -5.0

41. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 20% Improvement (ACR 20) Response at Week 52
Description: as for outcome 1
Time Frame: Baseline and Week 52
Population: The Apremilast participants as Randomized/Transitioned (AAR) Population; participants with a Baseline value and a Week 52 value are included.
  Reporting Groups
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo/Apremilast 20mg EE: Participants who received placebo twice daily up to Week 16 and were then transitioned to receive 20 mg apremilast twice daily.
- Placebo/Apremilast 20 mg XO: Participants who received placebo twice daily up to Week 24 and were then transitioned to receive 20 mg apremilast twice daily.
Arm/Group | Placebo/Apremilast 20mg EE | Placebo/Apremilast 20 mg XO | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 23 | 39 | 55 | 55
percentage of participants | 47.8 [26.8 to 69.4] | 51.3 [34.8 to 67.6] | 30.9 [19.1 to 44.8] | 38.2 [25.4 to 52.3]

42. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) at Week 52
Description: as for outcome 2
Time Frame: Baseline and Week 52
Population: The Apremilast participants as Randomized/Transitioned (AAR) Population; participants with a Baseline value and a Week 52 value are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo/Apremilast 20 mg XO: Participants who received placebo twice daily up to Week 24 and were then transitioned transitioned to receive 20 mg apremilast twice daily.
Arm/Group | Placebo/Apremilast 20mg EE | Placebo/Apremilast 20 mg XO | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 24 | 39 | 55 | 55
units on a scale | -0.219 (0.4287) | -0.192 (0.4728) | -0.155 (0.5501) | -0.277 (0.4281)

43. Secondary Outcome: Change From Baseline in the Medical Outcome Study Short Form 36-item (SF-36) Physical Functioning Domain at Week 52
Description: as for outcome 25
Time Frame: Baseline and Week 52
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Apremilast 20mg EE | Placebo/Apremilast 20 mg XO | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 24 | 39 | 55 | 55
units on a scale | 2.11 (6.959) | 3.50 (10.146) | 2.56 (9.978) | 5.23 (10.227)

44. Secondary Outcome: Change From Baseline in the Clinical Disease Activity Index (CDAI) at Week 52
Description: as for outcome 6
Time Frame: Baseline and Week 52
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Apremilast 20mg EE | Placebo/Apremilast 20 mg XO | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 23 | 39 | 55 | 55
units on a scale | -16.22 (8.722) | -20.70 (14.253) | -14.77 (14.220) | -17.68 (13.331)

45. Secondary Outcome: Percentage of Participants Who Achieve Low Disease Activity or Remission Based on the Clinical Disease Activity Index (CDAI) ≤ 10 at Week 52
Description: The Clinical Disease Activity Index (CDAI) is a composite index that is calculated as the sum of the:
  * 28 tender joint count (TJC),
  * 28 swollen joint count (SJC),
  * Subject's Global Assessment of Disease Activity measured on a 100 mm visual analog scale (VAS),, where 0 mm = lowest disease activity and 100 mm = highest;
  * Physician's Global Assessment of Disease Activity -measured on a 100 mm VAS, where 0 mm = lowest disease activity and 100 mm = highest.
  The CDAI score ranges from 0-76 where lower scores indicate less disease activity. The following thresholds of disease activity have been defined for the CDAI:
  Remission: ≤ 2.8; Low Disease Activity: > 2.8 and ≤ 10; Moderate Disease Activity: > 10 and ≤ 22; High Disease Activity: > 22
Time Frame: Baseline and Week 52
Population: as for outcome 42
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo/Apremilast 20mg EE | Placebo/Apremilast 20 mg XO | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 24 | 39 | 56 | 55
percentage of participants | 16.7 [4.7 to 37.4] | 41.0 [25.6 to 57.9] | 25.0 [14.4 to 38.4] | 27.3 [16.1 to 41.0]

46. Secondary Outcome: Change From Baseline in the Disease Activity Score 28 (DAS 28) Using CRP at Week 52
Description: The DAS28 measures the severity of disease at a specific time and is derived from the following variables:
  * 28 tender joint count (TJC28)
  * 28 swollen joint count (SJC28), which do not include the distal interphalangeal (DIP) joints, the hip joint, or the joints below the knee;
  * C-reactive protein (CRP)
  * Subject's global assessment of disease activity (SGA).
  DAS28 values range from 2.0 to 10.0 while higher values mean a higher disease activity.
  A DAS28 score higher than 5.1 indicates high disease activity, a DAS28 score less than 3.2 indicates low disease activity, and a DAS28 score less than 2.6 indicates clinical remission.
Time Frame: Baseline and Week 52
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Apremilast 20mg EE | Placebo/Apremilast 20 mg XO | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 23 | 39 | 54 | 55
units on a scale | -1.18 (0.717) | -1.68 (1.243) | -1.10 (1.290) | -1.38 (1.264)

47. Secondary Outcome: Percentage Change From Baseline in the Tender Joint Count at Week 52
Description: as for outcome 9
Time Frame: Baseline and Week 52
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo/Apremilast 20mg EE | Placebo/Apremilast 20 mg XO | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 24 | 40 | 56 | 55
percent change | -55.47 (24.072) | -62.70 (38.785) | -43.88 (38.728) | -54.03 (43.200)

48. Secondary Outcome: Percentage Change From Baseline in the Swollen Joint Count at Week 52
Description: as for outcome 10
Time Frame: Baseline and Week 52
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo/Apremilast 20mg EE | Placebo/Apremilast 20 mg XO | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 24 | 40 | 56 | 55
percent change | -59.40 (28.088) | -67.73 (42.431) | -57.31 (45.480) | -66.74 (30.277)

49. Secondary Outcome: Percentage Change From Baseline in the Subject Assessment of Pain at Week 52
Description: as for outcome 11
Time Frame: Baseline and Week 52
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo/Apremilast 20mg EE | Placebo/Apremilast 20 mg XO | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 24 | 39 | 55 | 55
percent change | 44.63 (184.396) [-33.23 to 122.50] | 15.78 (176.601) [-41.47 to 73.03] | -11.69 (42.608) [-23.20 to -0.17] | -3.73 (98.150) [-30.26 to 22.80]

50. Secondary Outcome: Percentage Change From Baseline in the Subject Global Assessment of Disease Activity at Week 52
Description: as for outcome 12
Time Frame: Baseline and Week 52
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Placebo/Apremilast 20 EE: Participants who received placebo twice daily up to Week 16 and were then transitioned to receive 20 mg apremilast twice daily.
- Placebo / Apremilast 20 mg XO: Participants who received placebo twice daily up to Week 24 and were then transitioned to receive 20 mg apremilast twice daily.
Arm/Group | Placebo/Apremilast 20 EE | Placebo / Apremilast 20 mg XO | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 24 | 39 | 55 | 55
percent change | 14.20 (76.243) | 33.31 (186.069) | -5.20 (73.593) | 8.22 (83.321)

51. Secondary Outcome: Percentage Change From Baseline in the Physician Global Assessment of Disease Activity at Week 52
Description: as for outcome 13
Time Frame: Baseline and Week 52
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo/Apremilast 20mg EE | Placebo/Apremilast 20 mg XO | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 23 | 40 | 56 | 55
percent change | -41.30 (35.683) | -49.10 (45.037) | -41.19 (47.417) | -44.85 (41.822)

52. Secondary Outcome: Percentage Change From Baseline in the Health Assessment Questionnaire - Disability Index (HAQ-DI) Score at Week 52
Description: as for outcome 2
Time Frame: Baseline and Week 52
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo/Apremilast 20mg EE | Placebo/Apremilast 20 mg XO | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 24 | 39 | 55 | 54
percent change | -13.32 (35.634) | -10.53 (49.600) | -8.20 (44.369) | -22.46 (31.856)

53. Secondary Outcome: Percentage Change From Baseline in the High Sensitivity C-Reactive Protein (CRP) at Week 52
Description: as for outcome 15
Time Frame: Baseline and Week 52
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo/Apremilast 20mg EE | Placebo/Apremilast 20 mg XO | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 23 | 40 | 55 | 55
percent change | 13.34 (90.641) | 82.14 (226.455) | 104.25 (210.138) | 79.33 (205.501)

54. Secondary Outcome: Percentage Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Week 52
Description: as for outcome 16
Time Frame: Baseline and Week 52
Population: The Apremilast Participants as Randomized/ Transitioned (AAR) Population; participants with a Baseline value and a Week 52 value are included.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo/Apremilast 20 EE | Placebo / Apremilast 20 mg XO | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 23 | 40 | 55 | 54
percent change | -6.28 (40.585) | 17.15 (244.497) | 4.83 (51.294) | -15.99 (53.892)

55. Secondary Outcome: Change From Baseline in the FACIT-Fatigue Scale Score at Week 52
Description: as for outcome 17
Time Frame: Baseline and Week 52
Population: as for outcome 54
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Apremilast 20mg EE | Placebo/Apremilast 20 mg XO | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 24 | 39 | 55 | 55
units on a scale | 3.50 (11.085) [22.1 to 63.4] | 3.18 (9.236) [44.6 to 76.6] | 2.87 (9.650) [32.0 to 59.4] | 3.47 (11.115) [27.0 to 54.1]

56. Secondary Outcome: Percentage of Participants Who Achieve an Improvement of ≥ 0.22 Units From Baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 52
Description: as for outcome 2
Time Frame: Baseline and Week 52
Population: as for outcome 42
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo/Apremilast 20mg EE | Placebo/Apremilast 20 mg XO | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 24 | 39 | 55 | 55
percentage of participants | 58.3 [36.6 to 77.9] | 43.6 [27.8 to 60.4] | 40.0 [27.0 to 54.1] | 58.2 [44.1 to 71.3]

57. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 50% Improvement (ACR 50) Response at Week 52
Description: as for outcome 23
Time Frame: Baseline and Week 52
Population: Apremilast participants as randomized during the apremilast exposure period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo/Apremilast 20 mg XO: .Participants who received placebo twice daily up to Week 24 and were then transitioned to receive 20 mg apremilast twice daily.
Arm/Group | Placebo/Apremilast 20mg EE | Placebo/Apremilast 20 mg XO | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 29 | 42 | 82 | 76
percentage of participants | 3.4 [0.1 to 17.8] | 11.9 [4.0 to 25.6] | 4.9 [1.3 to 12.0] | 5.3 [1.5 to 12.9]

58. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 70% Improvement (ACR 70) Response at Week 52
Description: Percentage of participants with an American College of Rheumatology 70% Improvement (ACR 70) response. A participant was a responder if the following 3 criteria for improvement from baseline were met:
  * ≥ 70% improvement in 68 tender joint count;
  * ≥ 70% improvement in 66 swollen joint count; and
  * ≥ 70% improvement in at least 3 of the 5 following parameters: Subject's assessment of pain (measured on a 100 mm visual analog scale [VAS]); Subject's global assessment of disease activity (measured on a 100 mm VAS); Physician's global assessment of disease activity (measured on a 100 mm VAS); Subject's self-assessment of physical function (Health Assessment Questionnaire - Disability Index ([HAQ-DI]); C-Reactive Protein
Time Frame: Baseline and Week 52
Population: Apremilast participants as randomized/transitioned (AAR Population); population consists of all participants who were randomized or transitioned to apremilast at any time during the study. Only those participants who had sufficient data for a definitive determination of response status at Week 52 are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo/Apremilast 20mg EE | Placebo/Apremilast 20 mg XO | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 24 | 40 | 56 | 55
percentage of participants | 0.0 [0.0 to 14.2] | 5.0 [0.6 to 16.9] | 7.1 [2.0 to 17.3] | 5.5 [1.1 to 15.1]

59. Secondary Outcome: Percentage of Participants Who Achieve an Improvement of at Least 4 Units From Baseline in the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) at Week 52
Description: as for outcome 39
Time Frame: Baseline and Week 52
Population: as for outcome 42
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo/Apremilast 20mg EE | Placebo/Apremilast 20 mg XO | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 24 | 39 | 55 | 55
percentage of participants | 41.7 [22.1 to 63.4] | 61.5 [44.6 to 76.6] | 45.5 [32.0 to 59.4] | 40.0 [27.0 to 54.1]

60. Secondary Outcome: Percentage of Participants Who Achieve the European League Against Rheumatism (EULAR) Response Criteria Using CRP at Week 52
Description: The EULAR response criteria classify each subject as a good, moderate or non-responder to treatment based on the degree of improvement from baseline and the level of disease activity at the endpoint. EULAR response is derived using the individual subject's DAS28 as the measure of severity of disease.
  Good or moderate response is defined as follows: Good response: DAS28 at the time point ≤ 3.2 and improvement from baseline > 1.2 Moderate response: DAS28 at the time point > 3.2 and improvement from baseline > 1.2, or DAS28 at the time point ≤ 5.1 and improvement from baseline > 0.6 and ≤ 1.2
Time Frame: Baseline and Week 52
Population: The Apremilast Participants as Randomized/ Transitioned (AAR) Population; only those participants who had sufficient data for a definitive determination of response status at Week 52 are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo/Apremilast 20mg EE | Placebo/Apremilast 20 mg XO | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 23 | 39 | 54 | 55
percentage of participants | 69.6 [47.0 to 86.8] | 82.1 [66.5 to 92.5] | 63.0 [48.7 to 75.7] | 65.5 [51.4 to 77.8]

61. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 20% Improvement (ACR 20) Response at Year 2
Description: Percentage of participants with an American College of Rheumatology 20% Improvement (ACR 20) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met:
  * ≥ 20% improvement in 68 tender joint count;
  * ≥ 20% improvement in 66 swollen joint count; and
  * ≥ 20% improvement in at least 3 of the 5 following parameters: Subject's assessment of pain (measured on a 100 mm visual analog scale [VAS]); Subject's global assessment of disease activity (measured on a 100 mm VAS); Physician's global assessment of disease activity (measured on a 100 mm VAS); Subject's self-assessment of physical function (Health Assessment Questionnaire - Disability Index ([HAQ-DI]); C-Reactive Protein.
  The study was terminated before the 2-year time point was reached due to lack of clinical efficacy.
Time Frame: Baseline and Year 2
Population: Analysis not performed.
Arm/Group | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 0 | 0

62. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) at Year 2
Description: The Health Assessment Questionnaire - Disability Index (HAQ-DI) is a patient-reported questionnaire consisting of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and usual activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task are summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. Negative mean changes from Baseline in the overall score indicate improvement in functional ability.
  The study was terminated before the 2-year time point was reached due to lack of clinical efficacy.
Time Frame: Baseline and Year 2
Population: Analysis not performed.
Arm/Group | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 0 | 0

63. Secondary Outcome: Change From Baseline in the Medical Outcome Study Short Form 36-item (SF-36) Physical Functioning Domain at Year 2
Description: The Medical Outcome Study Short Form 36-Item Health Survey, Version 2 (SF-36) was a self-administered instrument that measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). The concepts measured by the SF-36 are not specific to any age, disease, or treatment group, allowing comparison of relative burden of different diseases and the relative benefit of different treatments. Norm-based scores were used in analyses, calibrated so that 50 is the average score and the standard deviation equals 10. Higher scores indicate a higher level of functioning. The physical functioning domain assesses limitations in physical activities because of health problems. A positive change from baseline score indicates an improvement.
  The study was terminated before the 2-year time point was reached due to lack of clinical efficacy.
Time Frame: Baseline and Year 2
Population: Analysis not performed.
Arm/Group | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 0 | 0

64. Secondary Outcome: Change From Baseline in the Clinical Disease Activity Index (CDAI) at Year 2
Description: The Clinical Disease Activity Index (CDAI) is a composite index that is calculated as the sum of the:
  * 28 tender joint count (TJC),
  * 28 swollen joint count (SJC),
  * Subject's Global Assessment of Disease Activity measured on a 10 mm visual analog scale (VAS), where 0 mm = lowest disease activity and 10 mm = highest;
  * Physician's Global Assessment of Disease Activity -measured on a 10 mm VAS, where 0 mm = lowest disease activity and 10 mm = highest.
  The CDAI score ranges from 0-76 where lower scores indicate less disease activity. The following thresholds of disease activity have been defined for the CDAI:
  Remission: ≤ 2.8 Low Disease Activity: > 2.8 and ≤ 10 Moderate Disease Activity: > 10 and ≤ 22 High Disease Activity: > 22
  The study was terminated before the 2-year time point was reached due to lack of clinical efficacy.
Time Frame: Baseline and Year 2
Population: Analysis not performed.
Arm/Group | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 0 | 0

65. Secondary Outcome: Percentage of Participants Who Achieve Low Disease Activity or Remission Based on the Clinical Disease Activity Index (CDAI) ≤ 10 at Year 2
Description: as for outcome 64
Time Frame: Baseline and Year 2
Population: Analysis not performed.
Arm/Group | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 0 | 0

66. Secondary Outcome: Change From Baseline in Disease Activity Score 28 (DAS28) (Using C-Reactive Protein) (CRP) at Year 2
Description: The DAS 28 measures the severity of disease at a specific time and is derived from the following variables:
  * 28 tender joint count (TJC28)
  * 28 swollen joint count (SJC28), which do not include the distal interphalangeal (DIP) joints, the hip joint, or the joints below the knee;
  * C-reactive protein (CRP)
  * Subject's global assessment of disease activity (SGA ). A DAS28 score higher than 5.1 indicates high disease activity, a DAS28 score less than 3.2 indicates low disease activity, and a DAS28 score less than 2.6 indicates clinical remission.
  DAS28 values range from 2.0 to 10.0 while higher values mean a higher disease activity.
  The study was terminated before the 2-year time point was reached due to lack of clinical efficacy.
Time Frame: Baseline and Year 2
Population: Analysis not performed.
Arm/Group | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 0 | 0

67. Secondary Outcome: Percentage Change From Baseline in the Individual American College of Rheumatology Components at Year 2
Description: The Individual ACR Components were defined as follows:
  1. Tender Joint Count (out of 68 joints)
  2. Swollen Joint Count (out of 66 joints)
  3. Subject Assessment of Pain (0 to 100 mm VAS)
  4. Subject Global Assessment of Disease Activity (0 to 100 mm VAS)
  5. Physician Global Assessment of Disease Activity (0 to 100 mm VAS)
  6. HAQ-DI Score
  7. Acute Phase Reactant High Sensitivity C-Reactive Protein (hsCRP, mg/dL) Erythrocyte Sedimentation Rate (ESR)
  The study was terminated before the 2-year time point was reached due to lack of clinical efficacy.
Time Frame: Baseline and Year 2
Population: Analysis not performed.
Arm/Group | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 0 | 0

68. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy -Fatigue (FACIT-Fatigue) at Year 2
Description: The FACIT-Fatigue scale is a 13-item self-administered questionnaire that assesses both the physical and functional consequences of fatigue. Each question is answered on a 5-point scale, where 0 means "not at all," and 4 means "very much." The FACIT-Fatigue scale score ranges from 0 to 52, with higher scores denoting lower levels of fatigue.
  A positive change from baseline score indicates an improvement.
  The study was terminated before the 2-year time point was reached due to lack of clinical efficacy.
Time Frame: Baseline and Year 2
Population: Analysis not performed.
Arm/Group | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 0 | 0

69. Secondary Outcome: Percentage of Participants Who Achieve an Improvement of ≥ 0.22 Units From Baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI) at Year 2
Description: The Health Assessment Questionnaire - Disability Index (HAQ-DI) was a patient-reported questionnaire consisting of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and usual activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task are summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. Negative mean changes from Baseline in the overall score indicate improvement in functional ability.
  The study was terminated before the 2-year time point was reached due to lack of clinical efficacy.
Time Frame: Baseline and Year 2
Population: Analysis not performed.
Arm/Group | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 0 | 0

70. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 50% Improvement (ACR 50) Response at Year 2
Description: Percentage of participants with an American College of Rheumatology 50% Improvement (ACR 50) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met:
  * ≥ 50% improvement in 68 tender joint count;
  * ≥ 50% improvement in 66 swollen joint count; and
  * ≥ 50% improvement in at least 3 of the 5 following parameters: Subject's assessment of pain (measured on a 100 mm visual analog scale [VAS]); Subject's global assessment of disease activity (measured on a 100 mm VAS); Physician's global assessment of disease activity (measured on a 100 mm VAS); Subject's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [(HAQ-DI)]); C-Reactive Protein.
  The study was terminated before the 2-year time point was reached due to lack of clinical efficacy.
Time Frame: Baseline and Year 2
Population: Analysis not performed.
Arm/Group | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 0 | 0

71. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 70% Improvement (ACR 70) Response at Year 2
Description: Percentage of participants with an American College of Rheumatology 70% Improvement (ACR 70) response. A participant was a responder if the following 3 criteria for improvement from baseline were met:
  * ≥ 70% improvement in 68 tender joint count;
  * ≥ 70% improvement in 66 swollen joint count; and
  * ≥ 70% improvement in at least 3 of the 5 following parameters: Subject's assessment of pain (measured on a 100 mm visual analog scale [VAS]); Subject's global assessment of disease activity (measured on a 100 mm VAS); Physician's global assessment of disease activity (measured on a 100 mm VAS); Subject's self-assessment of physical function (Health Assessment Questionnaire - Disability Index ([HAQ-DI]); C-Reactive Protein
  The study was terminated before the 2-year time point was reached due to lack of clinical efficacy.
Time Frame: Baseline and Year 2
Population: Analysis not performed.
Arm/Group | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 0 | 0

72. Secondary Outcome: Percentage of Participants Who Achieve an Improvement of at Least 4 Units From Baseline in the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) at Year 2
Description: The FACIT-Fatigue scale was a 13-item self-administered questionnaire that assesses both the physical and functional consequences of fatigue. Each question is answered on a 5-point scale, where 0 means "not at all," and 4 means "very much." The FACIT-Fatigue scale score ranges from 0 to 52, with higher scores denoting lower levels of fatigue.
  The study was terminated before the 2-year time point was reached due to lack of clinical efficacy.
Time Frame: Baseline and Year 2
Population: Analysis not performed.
Arm/Group | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 0 | 0

73. Secondary Outcome: Percentage of Participants Who Achieve the European League Against Rheumatism (EULAR) Response Criteria Using CRP at Year 2
Description: EULAR response criteria classify each participant as a good, moderate or non-responder to treatment based on the degree of improvement from baseline and the level of disease activity at the endpoint. EULAR response is derived using the individual subject's DAS28 as the measure of severity of disease.
  Good or moderate response is defined as follows: Good response: DAS28 at the time point ≤ 3.2 and improvement from baseline > 1.2 Moderate response: DAS28 at the time point > 3.2 and improvement from baseline > 1.2, or DAS28 at the time point ≤ 5.1 and improvement from baseline > 0.6 and ≤ 1.2
  The study was terminated before the 2-year time point was reached due to lack of clinical efficacy.
Time Frame: Baseline and Year 2
Population: Analysis not performed.
Arm/Group | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All AEs were recorded by the Investigator from the time the participant signed the informed consent to 28 days after the last dose of investigational product.
Groups:
- Week 24: Placebo: Participants randomized to placebo tablets twice daily during the placebo-controlled phase. Includes data through Week 16 for participants who escaped early, and through Week 24 for all other participants.
- Week 24: Apremilast 20 mg: Participants randomized to receive 20 mg apremilast tablets twice daily during the 24-week placebo-controlled phase.
- Week 24: Apremilast 30 mg: Participants randomized to receive 30 mg apremilast tablets twice daily during the 24-week placebo-controlled phase.
- Study Termination: Apremilast 20 mg: Participants who received 20 mg apremilast, regardless of when the apremilast exposure started (at Week 0, 16, or 24), up until Study Termination.
- Study Termination: Apremilast 30 mg: Participants who received 30 mg apremilast, regardless of when the apremilast exposure started (at Week 0, 16, or 24), up until Study Termination.
Arm/Group | Week 24: Placebo | Week 24: Apremilast 20 mg | Week 24: Apremilast 30 mg | Study Termination: Apremilast 20 mg | Study Termination: Apremilast 30 mg
Serious Adverse Events (participants affected / at risk) | 1/79 | 6/82 | 4/76 | 16/153 | 7/76
Other Adverse Events (participants affected / at risk) | 15/79 | 26/82 | 23/76 | 49/153 | 29/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Week 24: Placebo (N=79) | Week 24: Apremilast 20 mg (N=82) | Week 24: Apremilast 30 mg (N=76) | Study Termination: Apremilast 20 mg (N=153) | Study Termination: Apremilast 30 mg (N=76)
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Staphylococcal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Costochondritis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Empyema (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Meningitis viral (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Mesothelioma malignant advanced (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Rheumatoid vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Foreign body reaction (General disorders) | 0 | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Pubis Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Cardiac congestive failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Week 24: Placebo (N=79) | Week 24: Apremilast 20 mg (N=82) | Week 24: Apremilast 30 mg (N=76) | Study Termination: Apremilast 20 mg (N=153) | Study Termination: Apremilast 30 mg (N=76)
Nasopharyngitis (Infections and infestations) | 4 | 6 | 3 | 11 | 6
Upper respiratory tract infecetion (Infections and infestations) | 2 | 3 | 5 | 9 | 7
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 4 | 4 | 4
Headache (Nervous system disorders) | 1 | 9 | 7 | 12 | 8
Hypertension (Vascular disorders) | 0 | 2 | 0 | 9 | 1
Nausea (Gastrointestinal disorders) | 6 | 7 | 10 | 13 | 10
Diarrhoea (Gastrointestinal disorders) | 2 | 7 | 6 | 14 | 6
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3 | 5 | 3 | 5
Vomiting (Gastrointestinal disorders) | 1 | 1 | 3 | 3 | 5

LIMITATIONS AND CAVEATS:
The study was terminated before the 2-year time point was reached due to lack of clinical efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 days. Investigator must delete confidential information before submission or defer publication to permit patent applications.